CLINICAL TRIAL: NCT03780959
Title: Safety, Population Pharmacokinetics, and Efficacy of Recombinant Human Tumor Necrosis Factor Receptor Fusion Protein (TNFR:Fc) in Children With Juvenile Rheumatoid Arthritis
Brief Title: Safety and Efficacy of Etanercept (Recombinant Human Tumor Necrosis Factor Receptor Fusion Protein [TNFR:Fc]) in Children With Juvenile Rheumatoid Arthritis (JRA)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20021616; 016.0016 (Other: Immunex Corporation)
Record Dates: First submitted 2018-12-18; First posted 2018-12-19 (Actual); Results first posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-06

CONDITIONS: Juvenile Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Etanercept/Placebo (Placebo Comparator): Participants received 0.4 mg/kg etanercept twice weekly for 90 days during Part 1. In Part 2 participants were randomized to receive placebo subcutaneous injection twice weekly for up to 4 months.
  Interventions: Drug: Etanercept; Drug: Placebo
- Etanercept/Etanercept (Experimental): Participants received 0.4 mg/kg etanercept twice weekly for 90 days during Part 1. In Part 2 participants were randomized to continue receiving etanercept twice weekly for up to 4 additional months.
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Administered twice weekly by subcutaneous injection
  Other Names: Enbrel; TNFR:Fc
Drug: Placebo — Administered twice weekly by subcutaneous injection
  Arms: Etanercept/Placebo

SUMMARY:
The primary objective of this study was to determine the efficacy of etanercept in children with polyarticular course JRA.

DETAILED DESCRIPTION:
This was a two-part study. In the first part of the study, all participants received open-label etanercept twice a week for 90 days. At the end of the 90 days, participants with disease response as defined by the JRA Definition of Improvement (DOI) using the JRA Core Set Criteria were randomized in part 2 of the study to receive placebo or continued administration of etanercept until either disease flare occurred or 4 months elapsed, whichever was earlier.

Participants who did not meet the DOI at day 90, participants who had disease flare during part 2 and participants who completed the blinded part of the study were eligible to receive open-label treatment with etanercept under protocol 16.0018 (NCT00357903).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of JRA by the American College of Rheumatology (ACR) criteria.
* Disease course must be polyarticular with disease duration long enough to have been given an adequate trial of non-steroidal anti-inflammatory drugs (NSAIDs) and low-dose methotrexate at a dose of at least 10 mg/m²/week
* Continuing active disease, defined as ≥ 5 swollen joints and ≥ 3 joints with limitation of motion accompanied by pain, tenderness or warmth.
* Disease refractory to methotrexate or intolerant of methotrexate.
* Have not received disease-modifying anti-rheumatic drugs (DMARDs) within 28 days prior to enrollment.
* Have not received methotrexate within 14 days prior to dosing of study drug.

Exclusion Criteria:

* Pregnant or nursing female
* Functional class IV by ACR criteria
* Unable to meet concomitant medication restrictions
* Intraarticular corticosteroid injection within 4 weeks prior to enrollment
* Clinically significant deviations from normal, defined as:

  * thrombocytopenia; platelet count < 100,000/cmm
  * leukopenia; total white cell count < 4000 cells/cmm
  * neutropenia; neutrophils < 1000 cells/cmm
  * hepatic transaminase levels > two times the upper limit of normal (ULN)
  * serum bilirubin > 2 times ULN
  * creatinine clearance < 90 mL/min/1.73 m² body surface area (BSA) and/or a glomerular filtration rate (GFR) < 90 mL/min/1.73 m² BSA.
  * known human immunodeficiency virus (HIV), hepatitis B surface antigen positivity, or hepatitis C positivity.
  * anti-double-stranded deoxyribonucleic acid (dsDNA) antibodies or anti-cardiolipin antibodies present.
* Previously received antibody to TNF, antibody to cluster of differentiation (CD)4, or diphtheria interleukin (IL)-2-fusion protein (DAB-IL-2)
* Participated in a study of an investigational drug or biologic requiring informed consent within 3 months prior to study entry.
* Any concurrent medical condition which would, in the investigator's opinion, compromise the patient's ability to tolerate the study drug or make the patient unable to cooperate with the protocol.
* History of or current psychiatric illness that would interfere with ability to comply with protocol requirements or informed consent.
* History or drug or alcohol abuse that would interfere with ability to comply with protocol requirements

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 69 (Actual)
Dates: Start 1997-05-01 (Actual); Primary Completion 1998-07-08 (Actual); Study Completion 1998-07-08 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 9 sites in the United States and Canada. The study consisted of an open-label treatment period (part 1) where all participants received 0.4 mg etanercept twice weekly for 3 months, followed by a randomized double-blind treatment period (part 2).
Pre-assignment Details: At the end of part 1 participants with disease response were randomized to part 2, with stratification according to study center and number of active joints (≤ 2 vs. > 2) at the end of month 3.
Groups:
- Part 1: Etanercept 0.4 mg/kg: Participants received 0.4 mg/kg etanercept twice weekly for 90 days during Part 1.
- Part 2: Placebo: In Part 2 participants were randomized to receive placebo subcutaneous injection twice weekly for up to 4 months.
- Part 2: Etanercept 0.4 mg/kg: In Part 2 participants were randomized to continue receiving 0.4 mg/kg etanercept twice weekly for up to 4 additional months.
Period: Part 1
Arm/Group | Part 1: Etanercept 0.4 mg/kg | Part 2: Placebo | Part 2: Etanercept 0.4 mg/kg
Started | 69 | 0 | 0
Completed | 64 | 0 | 0
Not Completed | 5 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Withdrawal by Parent/Guardian | 1 | 0 | 0
Not completed — Response Status | 2 | 0 | 0
Period: Part 2
Arm/Group | Part 1: Etanercept 0.4 mg/kg | Part 2: Placebo | Part 2: Etanercept 0.4 mg/kg
Started (Participants who met response criteria at day 90) | 0 | 26 | 25
Completed | 0 | 7 | 19
Not Completed | 0 | 19 | 6
Not completed — Withdrawal by Parent/Guardian | 0 | 1 | 0
Not completed — Response Status | 0 | 18 | 6

BASELINE CHARACTERISTICS:
Population: Baseline data are included for all enrolled participants in part 1 (69) and all participants who randomized in part 2 (51).
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Etanercept 0.4 mg/kg | Part 2: Placebo | Part 2: Etanercept 0.4 mg/kg | Total
Number analyzed (Participants) | 69 | 26 | 25 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Part 1 and Part 2 baseline data are reported separately since Part 2 participants represent a subset of Part 1.
  years
    Part 1: number analyzed (Participants) | 69 | 0 | 0 | 69
    Part 1 | 10.5 (3.9) |  |  | 10.5 (3.9)
    Part 2: number analyzed (Participants) | 0 | 26 | 25 | 51
    Part 2 |  | 12.2 (3.5) | 8.9 (3.7) | 10.6 (3.9)
Age, Customized [Count of Participants; unit: Participants] — Population: Part 1 and Part 2 baseline data are reported separately since Part 2 participants represent a subset of Part 1.
  Participants
    Part 1: number analyzed (Participants) | 69 | 0 | 0 | 69
    Part 1: 4 - 8 years | 25 |  |  | 25
    Part 1: 9 - 12 years | 14 |  |  | 14
    Part 1: 13 - 17 years | 30 |  |  | 30
    Part 2: number analyzed (Participants) | 0 | 26 | 25 | 51
    Part 2: 4 - 8 years |  | 5 | 13 | 18
    Part 2: 9 - 12 years |  | 4 | 5 | 9
    Part 2: 13 - 17 years |  | 17 | 7 | 24
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Part 1 and Part 2 baseline data are reported separately since Part 2 participants represent a subset of Part 1.
  Participants
    Part 1: number analyzed (Participants) | 69 | 0 | 0 | 69
    Part 1: Female | 43 |  |  | 43
    Part 1: Male | 26 |  |  | 26
    Part 2: number analyzed (Participants) | 0 | 26 | 25 | 51
    Part 2: Female |  | 15 | 19 | 34
    Part 2: Male |  | 11 | 6 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Part 1 and Part 2 baseline data are reported separately since Part 2 participants represent a subset of Part 1.
  Participants
    Part 1: number analyzed (Participants) | 69 | 0 | 0 | 69
    Part 1: Black | 6 |  |  | 6
    Part 1: White | 52 |  |  | 52
    Part 1: Asian | 1 |  |  | 1
    Part 1: Hispanic | 9 |  |  | 9
    Part 1: Native American | 1 |  |  | 1
    Part 2: number analyzed (Participants) | 0 | 26 | 25 | 51
    Part 2: Black |  | 1 | 3 | 4
    Part 2: White |  | 23 | 14 | 37
    Part 2: Asian |  | 0 | 1 | 1
    Part 2: Hispanic |  | 2 | 6 | 8
    Part 2: Native American |  | 0 | 1 | 1
Type of Onset of Juvenile Rheumatoid Arthritis (JRA) [Count of Participants; unit: Participants] — Onset type is determined by manifestations during the first 6 months of disease.
  Pauciarticular JRA: Arthritis in 4 or fewer joints during the first 6 months of disease.
  Polyarticular JRA: Arthritis in 5 or more joints during the first 6 months of disease.
  Systemic onset JRA: Arthritis with persistent intermittent fever with or without rheumatoid rash or other organ involvement. Population: Part 1 and Part 2 baseline data are reported separately since Part 2 participants represent a subset of Part 1.
  Participants
    Part 1: number analyzed (Participants) | 69 | 0 | 0 | 69
    Part 1: Pauciarticular | 7 |  |  | 7
    Part 1: Polyarticular | 40 |  |  | 40
    Part 1: Systemic | 22 |  |  | 22
    Part 2: number analyzed (Participants) | 0 | 26 | 25 | 51
    Part 2: Pauciarticular |  | 1 | 2 | 3
    Part 2: Polyarticular |  | 17 | 14 | 31
    Part 2: Systemic |  | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Disease Flare in Part 2
Description: Disease flare was defined as a 30% or greater worsening in three of the six JRA Core Set Criteria and ≥ 30% improvement in one or less of the six JRA Core Set Criteria compared to day 90 and a minimum of two active joints (joints with swelling or limitation of movement plus pain and/or tenderness).
  The JRA Core Set criteria consisted of:
  * Physician global assessment of disease severity assessed on a visual analog scale (VAS) from 0 (asymptomatic) to 10 (severe symptoms);
  * Patient/parent global assessment of overall well-being assesses on a VAS from 0 (asymptomatic) to 10 (severe symptoms);
  * Number of active joints;
  * Number of joints with limitation of motion (LOM) and with pain, tenderness, or both;
  * Childhood Health Assessment Questionnaire (CHAQ) disability domain;
  * Erythrocyte sedimentation rate (ESR).
Time Frame: End of part 1 (day 90) and months 4 to 7
Population: All randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: Placebo | Part 2: Etanercept 0.4 mg/kg
Number analyzed (Participants) | 26 | 25
percentage of participants | 81 | 28
Statistical Analysis 1: Comparison: Part 2: Placebo vs Part 2: Etanercept 0.4 mg/kg; Test type: Superiority; p = 0.0030, Mantel Haenszel; Stratified by study center and the number of active joints at randomization

2. Secondary Outcome: Time to Flare in Part 2
Description: The time from day 90 to flare. Participants who withdrew without flare were censored at the time of withdrawal.
Time Frame: Months 4 to 7
Population: All randomized participants
Measure: Median (Full Range); unit: days
Arm/Group | Part 2: Placebo | Part 2: Etanercept 0.4 mg/kg
Number analyzed (Participants) | 26 | 25
days | 28.0 [6 to 123] | 116.0 [28 to 127]
Statistical Analysis 1: Comparison: Part 2: Placebo vs Part 2: Etanercept 0.4 mg/kg; Test type: Superiority; p = 0.0001, Log Rank

3. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: Part 1: 90 days (months 1-3) plus 30 days for participants who were not randomized into part 2. Part 2: From first dose of randomized treatment to 30 days after last dose (150 days; months 4-8).
Population: All participants who received at least one dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Etanercept 0.4 mg/kg | Part 2: Placebo | Part 2: Etanercept 0.4 mg/kg
Number analyzed (Participants) | 69 | 26 | 25
Participants
  Noninfectious adverse events | 51 | 9 | 13
  Injection site reactions | 27 | 1 | 1
  Infections | 43 | 8 | 15
  Serious adverse events | 1 | 0 | 1
  Deaths | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Part 1: 90 days (months 1-3) plus 30 days for participants who were not randomized into part 2. Part 2: From first dose of randomized treatment to 30 days after last dose (150 days; months 4-8).
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Part 2: Placebo: n Part 2 participants were randomized to receive placebo subcutaneous injection twice weekly for up to 4 months.
Arm/Group | Part 1: Etanercept 0.4 mg/kg | Part 2: Placebo | Part 2: Etanercept 0.4 mg/kg
Serious Adverse Events (participants affected / at risk) | 1/69 | 0/26 | 1/25
Other Adverse Events (participants affected / at risk) | 59/69 | 12/26 | 19/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Etanercept 0.4 mg/kg (N=69) | Part 2: Placebo (N=26) | Part 2: Etanercept 0.4 mg/kg (N=25)
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Etanercept 0.4 mg/kg (N=69) | Part 2: Placebo (N=26) | Part 2: Etanercept 0.4 mg/kg (N=25)
Abdominal pain upper (Gastrointestinal disorders) | 7 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 2
Nausea (Gastrointestinal disorders) | 7 | 0 | 2
Vomiting (Gastrointestinal disorders) | 10 | 0 | 3
Fatigue (General disorders) | 4 | 1 | 1
Injection site erythema (General disorders) | 23 | 1 | 0
Injection site pain (General disorders) | 10 | 1 | 0
Injection site pruritus (General disorders) | 13 | 1 | 0
Injection site swelling (General disorders) | 13 | 1 | 1
Pyrexia (General disorders) | 2 | 0 | 2
Ear infection (Infections and infestations) | 6 | 2 | 1
Gastroenteritis (Infections and infestations) | 5 | 1 | 3
Influenza (Infections and infestations) | 2 | 2 | 2
Pharyngitis (Infections and infestations) | 10 | 0 | 3
Tinea pedis (Infections and infestations) | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 24 | 4 | 10
Headache (Nervous system disorders) | 14 | 3 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 5 | 2 | 0
Vasculitic rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to1 review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.